CLINICAL TRIAL: NCT03150732
Title: Comparison of Systemic Nalbuphine Versus Intravenous Regional Anesthesia
Brief Title: Systemic Nalbuphine Versus Intravenous Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bakri, Professor of anesthesia & ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 000087273
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systemic nalbuphine group (Active Comparator): 53 patients will receive nalbuphine systemically
  Interventions: Drug: Systemic nalbuphine
- Local nalbuphine group (Active Comparator): 53 patients will receive nalbuphine with local intravenous regional anesthesia (IVRA)
  Interventions: Drug: Local nalbuphine

INTERVENTIONS:
Drug: Systemic nalbuphine — Patients will receive systemic nalbuphine 10 mg
  Arms: Systemic nalbuphine group
Drug: Local nalbuphine — Patients will receive local nalbuphine 10 mg
  Arms: Local nalbuphine group

SUMMARY:
Comparison of systemic nalbuphine versus intravenous regional anesthesia in patients undergoing hand surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective unilateral hand surgery.

Exclusion Criteria:

* Patient refusal.
* Allergy to study medications
* Body mass index > 35 kg/ m2
* Patients with sickle cell or Reynaud diseases
* Patients with a history of psychiatric illness or on chronic opioids

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative Analgesia | Postoperative 24 hours
  minutes

SECONDARY OUTCOMES:
Diclofenac analgesic consumption | Postoperative 24 hours
  mg
Cortisol level | Preoperative and at 4 hours after skin incision
  Level of cortisone in blood (nmol/L)
Severity of postoperative Pain | Postoperative 24 hours
  Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed H Bakri, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No